CLINICAL TRIAL: NCT05688553
Title: The Effects of Using Flexi-bar for Balance and Strength Training on the Balance and Muscle in Community-Dwelling Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-E(I)-20220165
Record Dates: First submitted 2022-09-23; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-11

CONDITIONS: Flexi-bar; Vibration; Balance Training; Community-dwelling; Community Older; Strength Training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexi-bar group (Experimental)
  Interventions: Device: Flexi-bar
- balance and strength group (Active Comparator)
  Interventions: Other: balance and strength training

INTERVENTIONS:
Device: Flexi-bar — two groups, experimental group intervention Flexi-bar with balance and strength training
  Arms: Flexi-bar group
Other: balance and strength training — the control group intervention only balance and strength training
  Arms: balance and strength group

SUMMARY:
Aging of the neuromuscular system may lead to an increased risk of falls in older adults. There are external and internal factors for falls, and lower limb muscle strength and balance are important internal factors for falls in the elderly. And can be improved through exercise. Therefore, an important interventional goal in interventional exercises to prevent falls in the elderly is to promote balance and increase lower extremity muscle strength.

Flexi-bar is a device that provides vibration stimulation. Studies have shown that a 5Hz frequency can be generated when shaken and transmitted to the whole body. Flexi bar is now widely used in fitness centers or rehabilitation therapy to improve muscle strength and balance. Vibration activates the tonic reflex, enhances the excitability of alpha and gamma motor neurons and enhances motor unit synchronization, and this active vibration training helps increase muscle coordination as it induces the tonic reflex and stimulates the proprioception of the joint Feelings, these physiological changes can lead to more effective proprioceptive feedback that improves balance. And because the vibration causes the agonist and antagonist muscles to contract alternately to regulate the instability during the movement. In recreational athletes, the use of a flexi bar in a single-legged position can effectively induce lower extremity muscle activation.

A 12-week combination of balance and strength training in older adults has been shown to be effective in reducing the risk of falls in older adults in previous studies.

Since the effect of adding Flexi bar on the basis of balance and strength training is unknown, the purpose of this study was to investigate the experimental group and the control group with the same exercise posture and training time, Flexi bar + BST Is it better for the balance and muscle strength of the elderly than simple BST?

ELIGIBILITY:
Inclusion Criteria:

•Elderly people aged 65 to 85 in the community who can move on their own without the need for support from others.

Exclusion Criteria:

* Vulnerable groups: those who lack sufficient decision-making ability due to age, intellectual or physical (physiological) status, or who are vulnerable to undue influence, coercion, or inability to make decisions of free will due to their environment, identity, or socioeconomic status, People living in nursing homes and racially disadvantaged groups, etc.
* Have been diagnosed with mental illness and cognitive impairment
* Those who have had severe cardiovascular-related diseases such as unstable angina pectoris, acute myocardial infarction and are not suitable for vigorous exercise
* Those with a history of epilepsy
* Those with severe pain in the lower extremity joints during the pre-test and unable to complete the above-mentioned lower extremity muscle strength or balance test.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline gait and balance at 12 weeks | baseline , up to 12 weeks( post test)
  Functional gait assessment
change from baseline dynamic balance at 12 weeks | baseline , up to 12 weeks( post test)
  Y-Balance Test
change from baseline balance at 12 weeks | baseline , up to 12 weeks( post test)
  Mini-Balance Evaluation Systems Test

SECONDARY OUTCOMES:
change from baseline lower strength at 12 weeks (1) | baseline , up to 12 weeks( post test)
  Chair standing test
change from baseline lower strength at 12 weeks(2) | baseline , up to 12 weeks( post test)
  hand held dynamometer
change from baseline ankle plantar flexor strength at 12 weeks | baseline , up to 12 weeks( post test)
  ankle plantar flexion test

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiang Li Activity Center, Kaohsiung City, Taiwan